CLINICAL TRIAL: NCT04351555
Title: A Phase III, Randomised, Controlled, Multi-center, 3-Arm Study of Neoadjuvant Osimertinib as Monotherapy or in Combination With Chemotherapy Versus Standard of Care Chemotherapy Alone for the Treatment of Patients With Epidermal Growth Factor Receptor Mutation Positive, Resectable Non-small Cell Lung Cancer
Brief Title: A Study of Osimertinib With or Without Chemotherapy Versus Chemotherapy Alone as Neoadjuvant Therapy for Patients With EGFRm Positive Resectable Non-Small Cell Lung Cancer
Acronym: NeoADAURA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D516AC00001; 2022-502606-33-00 (Registry Identifier: CTIS (EU)); 2020-000058-89 (EudraCT Number)
Record Dates: First submitted 2020-04-01; First posted 2020-04-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Resectable; NSCLC; Osimertinib; EGFRm Positive; Neoadjuvant; Adjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The two arms with SoC chemotherapy (placebo plus chemotherapy versus osimertinib plus chemotherapy) will be double-blinded and placebo-controlled.
  Osimertinib monotherapy arm will be open label, sponsor-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Placebo with platinum-based chemotherapy (Placebo Comparator): Placebo plus investigator's choice of platinum-based standard of care chemotherapy (pemetrexed/carboplatin or pemetrexed/cisplatin)
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Placebo; Drug: Pemetrexed
- Arm 2: Osimertinib with platinum-based chemotherapy (Experimental): Osimertinib 80 mg QD (Dose may be reduced to 40 mg QD at the discretion of the investigator) plus investigator's choice of platinum-based standard of care chemotherapy (pemetrexed/carboplatin or pemetrexed/cisplatin)
  Interventions: Drug: Osimertinib; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Arm 3: Osimertinib monotherapy (Experimental): Osimertinib 80 mg QD (Dose may be reduced to 40 mg QD at the discretion of the investigator)
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Oral
  Other Names: AZD9291; TAGRISSO
  Arms: Arm 2: Osimertinib with platinum-based chemotherapy; Arm 3: Osimertinib monotherapy
Drug: Cisplatin — Cisplatin (75mg/m2) to be administered with pemetrexed on Day 1 of every 3-week cycle for 3 cycles.
  Arms: Arm 1: Placebo with platinum-based chemotherapy; Arm 2: Osimertinib with platinum-based chemotherapy
Drug: Carboplatin — Carboplatin (AUC5) to be administered with pemetrexed on Day 1 of every 3-week cycle for 3 cycles
  Arms: Arm 1: Placebo with platinum-based chemotherapy; Arm 2: Osimertinib with platinum-based chemotherapy
Drug: Placebo — Oral
  Arms: Arm 1: Placebo with platinum-based chemotherapy
Drug: Pemetrexed — Pemetrexed (500 mg/m2) to be administered with cisplatin or carboplatin on Day 1 of every 3-week cycle for 3 cycles
  Arms: Arm 1: Placebo with platinum-based chemotherapy; Arm 2: Osimertinib with platinum-based chemotherapy

SUMMARY:
This is a Phase III, randomised, controlled, 3-arm, multi-centre study of neoadjuvant osimertinib as monotherapy or in combination with chemotherapy, versus SoC chemotherapy alone, for the treatment of patients with resectable EGFRm Non-Small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age. For patients aged <20 years and enrolled in Japan, a written informed consent should be obtained from the patient and his or her legally acceptable representative
* Histologically or cytologically documented non-squamous NSCLC with completely resectable (Stage II - IIIB N2) disease (according to Version 8 of the IASLC Cancer Staging Manual [IASLC Staging Manual in Thoracic Oncology 2016]).
* Complete surgical resection of the primary NSCLC must be deemed achievable, as assessed by a MDT evaluation (which should include a thoracic surgeon, specialised in oncologic procedures).
* Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1 at enrolment, with no deterioration over the previous 2 weeks prior to baseline or day of first dosing
* A tumour which harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations (eg., T790M, G719X, Exon20 insertions, S7681 and L861Q).

Exclusion Criteria:

* Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* History of another primary malignancy (including any known or suspected synchronous primary lung cancer), except for the following: Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of investigational product (IP) and of low potential risk for recurrence; Adequately treated non-melanoma skin cancer or lentigo malignancy without evidence of disease; Adequately treated carcinoma in situ without evidence of disease; Any synchronous Stage IA primary lung cancer that is ≤2 cm and planned to be resected during surgery for the Stage II to IIIB N2 lung tumour.
* Patients who have pre-operative radiotherapy treatment as part of their care plan
* Mixed small cell and NSCLC histology
* Stages I, IIIB N3, IIIC, IVA, and IVB NSCLC
* T4 tumours infiltrating the great vessels, the carina, the trachea, the oesophagus, the heart, and/or the vertebral body; and/or any bulky N2 disease.
* Patients who are candidates to undergo only segmentectomies or wedge resections
* Prior treatment with any systemic anti-cancer therapy for NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug
* Prior treatment with EGFR-TKI therapy
* Current use of (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of cytochrome P450 (CYP) 3A4 (at least 3 weeks prior)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2029-06-13 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | From date of randomization to an average of 12 weeks after the first dose
  Defined as ≤10% residual cancer cells in the main tumour, as assessed per central pathology laboratory post-surgery

SECONDARY OUTCOMES:
Pathological complete response (pCR) | From date of randomization to an average of 12 weeks after the first dose
  Defined as absence of any viable cancer cells in the dissected tumour samples, including the main tumour, lymph nodes, and margins as assessed per central pathology laboratory post-surgery
Event-free survival (EFS) | From date of randomization up to approximately 5.5 years after the last patient is randomized
  An event is defined as documented disease progression that precludes surgery or prevents completion of definitive surgery; recurrence or a new lesion, local or distant (a new primary malignancy, confirmed by pathology if clinically feasible, is not considered to be an EFS event); death due to any cause
Overall Survival (OS) | From date of randomization up to approximately 5.5 years after the last patient is randomized
  OS will be defined as the time from the date of randomisation until death due to any cause
Disease free survival (DFS) | From date of randomization up to approximately 5.5 years after the last patient is randomized
  DFS is defined as the time from the date of surgery until the first date of disease recurrence (local or distant) or date of death due to any cause, whichever occurs first.
Downstaging | From date of randomization to an average of 12 weeks after the first dose
  Measured using pathologic mediastinal lymph node evaluation
Difference between treatment arms in change from baseline in EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 items) | From date of randomization up to approximately 5.5 years after the last patient is randomized
  Assess disease-related symptoms, functioning, and global health status/quality-of-life in patients
Concordance of EGFRm status between tumour tissue DNA and patient-matched plasma-derived ctDNA | Baseline
Corcordance of EGFR mutation status between the local and central cobas EGFR mutation test results from baseline tumour samples | Baseline
PK plasma concentrations of osimertinib | From the pre-dose of Cycle 2 to post-dose of Cycle 3 (each cycle is 21 days)
Difference between treatment arms in change from baseline in EORTC QLQ-LC13 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 items) | From date of randomization up to approximately 5.5 years after the last patient is randomized
  Assess lung cancer-associated symptoms and side effects from conventional chemotherapy and radiotherapy

OTHER OUTCOMES:
Cure rate | From the surgery until 5 years after surgery
  The cure rate is defined as the percentage of people in this study who are still alive and disease free for a certain period of time after they finished the surgery. Here 5-year landmark cure rate will be calculated in the same time as OS analysis.
Number of adverse events as assessed by CTCAE 5.0 and other clinical variables for safety and tolerability profile of neoadjuvant osimertinib as monotherapy or in combination with chemotherapy prior to surgery compared with chemotherapy alone | From the time of enrollment to either 28-days after the last dose of last study treatment for patients who do not undergo surgery, or 90-days post-surgery
  Other clinical variables include deaths, laboratory data, vital signs (pulse and BP), ECG, LVEF, ECOG performance status, and ophthalmologic assessment
MPR using plasma-derived circulating-free tumour DNA (ctDNA) | From date of randomization to an average of 12 weeks after the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Chaft, MD, Principal Investigator — Memorial Sloan Kettering, USA; Masahiro Tsuboi, MD, Principal Investigator — National Cancer Center Hospital East, Japan; Walter Weder, MD, Principal Investigator — Thoraxchirurgie Bethanien, Switzerland
Locations (130):
- United States (12):
  - Research Site, Duarte, California
  - Research Site, Irvine, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, Santa Rosa, California
  - Research Site, Boston, Massachusetts
  - Research Site, Lebanon, New Hampshire
  - Research Site, Commack, New York
  - Research Site, New York, New York
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Seattle, Washington
- Austria (2):
  - Research Site, Graz
  - Research Site, Vienna
- Brazil (9):
  - Research Site, Barretos
  - Research Site, Fortaleza
  - Research Site, Jaú
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, Santa Maria
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (3):
  - Research Site, Panagyurishte
  - Research Site, Pleven
  - Research Site, Sofia
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Chile (2):
  - Research Site, Las Condes
  - Research Site, Santiago
- China (17):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Kunming
  - Research Site, Nanchang
  - Research Site, Nantong
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Ürümqi
  - Research Site, Wanzhou
  - Research Site, Wenzhou
  - Research Site, Xiamen
  - Research Site, Yangzhou
- France (2):
  - Research Site, Avignon
  - Research Site, Bordeaux
- Germany (10):
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Cologne
  - Research Site, Esslingen a.N.
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Georgsmarienhütte
  - Research Site, Halle
  - Research Site, Oldenburg
  - Research Site, Würzburg
- India (4):
  - Research Site, Mumbai
  - Research Site, Namakkal
  - Research Site, New Delhi
  - Research Site, Varanasi
- Israel (6):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (7):
  - Research Site, Bari
  - Research Site, Florence
  - Research Site, Monza
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Rozzano
  - Research Site, Varese
- Japan (15):
  - Research Site, Akashi-shi
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Hiroshima
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Kyoto
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sakaishi
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Mexico (3):
  - Research Site, Aguascalientes
  - Research Site, D.F
  - Research Site, Mexico City
- Peru (2):
  - Research Site, La Libertad
  - Research Site, Lima
- Research Site, Olsztyn, Poland
- Russia (7):
  - Research Site, Kazan'
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Obninsk
  - Research Site, Perm
  - Research Site, Saint Petersburg
- South Korea (5):
  - Research Site, Daegu
  - Research Site, Hwasun-gun
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Yangsan
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
- Switzerland (2):
  - Research Site, Winterthur
  - Research Site, Zurich
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
  - Research Site, Pathum Thani
  - Research Site, Phisanulok
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Malatya
- United Kingdom (2):
  - Research Site, Birmingham
  - Research Site, Liverpool
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] He J, Tsuboi M, Weder W, Chen KN, Hochmair MJ, Shih JY, Lee SY, Lee KY, Nhung NV, Saeteng S, Liu L, Xing L, Gia NH, Murakami S, Han Y, Saavedra MP, Yoon SH, Teixeira CHA, Escriu C, Martinez-Marti A, Blakely CM, Yatabe Y, Dacic S, Rukazenkov Y, Huang X, Dayal A, Chaft JE; NeoADAURA Investigators. Neoadjuvant Osimertinib for Resectable EGFR-Mutated Non-Small Cell Lung Cancer. J Clin Oncol. 2025 Sep 10;43(26):2875-2887. doi: 10.1200/JCO-25-00883. Epub 2025 Jun 2. PMID 40454705
- [Derived] Murat-Onana ML, Ramalingam SS, Janne PA, Gray JE, Ahn MJ, John T, Yatabe Y, Huang X, Rukazenkov Y, Javey M, Brown H, Li-Sucholeiki X. EGFR mutation testing across the osimertinib clinical program. Lung Cancer. 2025 Jun;204:108549. doi: 10.1016/j.lungcan.2025.108549. Epub 2025 Apr 18. PMID 40311309
- [Derived] Lee JB, Choi SJ, Shim HS, Park BJ, Lee CY, Sudhaman S, Velichko S, Hong MH, Cho BC, Lim SM. Neoadjuvant and Adjuvant Osimertinib in Stage IA to IIIA, EGFR-Mutant NSCLC (NORA). J Thorac Oncol. 2025 May;20(5):641-650. doi: 10.1016/j.jtho.2024.12.023. Epub 2024 Dec 26. PMID 39732365
- [Derived] Tsuboi M, Weder W, Escriu C, Blakely C, He J, Dacic S, Yatabe Y, Zeng L, Walding A, Chaft JE. Neoadjuvant osimertinib with/without chemotherapy versus chemotherapy alone for EGFR-mutated resectable non-small-cell lung cancer: NeoADAURA. Future Oncol. 2021 Nov;17(31):4045-4055. doi: 10.2217/fon-2021-0549. Epub 2021 Jul 19. PMID 34278827